CLINICAL TRIAL: NCT03271736
Title: Effects of Rhythmic Auditory Cueing on Stepping in Place in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HsiuYun Chang (Other)
Responsible Party: Sponsor-Investigator, HsiuYun Chang, Principal Investigator, National Taiwan University
Organization: National Taiwan University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201609085RINA
Record Dates: First submitted 2017-08-06; First posted 2017-09-05 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Auditory cues; step in place; transcranial magnetic stimulation; cortical excitability
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freezer (Experimental): All the subjects received 2 experiments. 2 experiments contain 20 mins stepping-in-place exercise and pre-/post assessments. The difference between 2 experiments is the application of auditory cues. One of the 2 experiment includes stepping-in-place exercise with auditory cues from the metronome (Stepping-in-place exercise with external auditory cues), in the other experiment we ask the subjects to follow their internal rhythm without external auditory cues (Stepping-in-place exercise without external auditory cues). Transcranial magnetic stimulation (TMS) is applied before and after the stepping-in-place exercise.
  Interventions: Behavioral: Stepping-in-place exercise with external auditory cues; Device: Transcranial magnetic stimulation (TMS)
- Non-freezer (Experimental): All the subjects received 2 experiments. 2 experiments contain 20 mins stepping-in-place exercise and pre-/post assessments. The difference between 2 experiments is the application of auditory cues. One of the 2 experiment includes stepping-in-place exercise with auditory cues from the metronome (Stepping-in-place exercise with external auditory cues), in the other experiment we ask the subjects to follow their internal rhythm without external auditory cues (Stepping-in-place exercise without external auditory cues). Transcranial magnetic stimulation (TMS) is applied before and after the stepping-in-place exercise.
  Interventions: Behavioral: Stepping-in-place exercise with external auditory cues; Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Behavioral: Stepping-in-place exercise with external auditory cues — The stepping-in-place exercise includes 10-session training. In each session, subjects are asked for stepping for 50 steps. In auditory cued condition, the cued frequency is set at 110% of the usual walking cadence. While in non-cued condition, we ask the subjects to step according to their own internal rhythm.
  Other Names: Stepping-in-place exercise without external auditory cues
Device: Transcranial magnetic stimulation (TMS) — TMS is used to assess the cortical excitability of the motor cortex. The stimulation intensity is set at 130% of the motor threshold in single-pulse condition. In paired-pulse condition, the first stimulus is set at 80% of the motor threshold and the second stimulus is set at 130% of the motor threshold.

SUMMARY:
Patients with Parkinson's disease have internal rhythm dysfunction, which may affect the rhythmic movements such as walking. Poor regularity of the rhythmic movement may lead to freezing of gait. This study will apply rhythmic auditory cues on the stepping-in-place training and the investigators will examine if the behavior and neuroelectrophysiology would change after auditory cueing training. The investigators hypothesize the variation of rhythmic movements such as walking and stepping-in-place will be reduced, and the cortical excitability would be modulated after training.

DETAILED DESCRIPTION:
Parkinson's disease is a common neurodegenerative disease and movement disorder. Due to the degeneration of basal ganglia, patients with Parkinson's disease also demonstrate internal rhythm dysfunction, thus will lead to difficulty in rhythmic movements such as ambulation. For improving the rhythmic movement problem, auditory cues are often used in clinical setting and shows benefits in ambulation and freezing problems. Previous studies often use finger tapping test and ambulation to assess the rhythmic movement problem. No study uses stepping in place movements as a test to examine rhythmic problem. Little study investigates the effects of auditory cues on brain cortical excitability. In this cross-over study, participants will receive 2 times of training include stepping-in-place exercise with and without auditory cues in random orders. Auditory cues are given via the metronome. There is one-week wash-out period between two trainings. Movement tests such as walking and stepping-in-place and transcranial magnetic stimulation (TMS) are carried out before and after each training.

The investigators hypothesize the variation of rhythmic movements such as walking and stepping-in-place will be reduced more, and the cortical excitability would be modulated after the training with auditory cues, comparing with the other training without auditory cues.

ELIGIBILITY:
[Patients with Parkinson's disease]

Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease
* No hearing impairment
* Able to walk independently for at least 10m
* Able to follow command (MMSE >=24)

[Healthy subjects]

* No hearing impairment
* Able to walk independently for at least 10m
* Able to follow command (MMSE >=24)

Exclusion Criteria:

* With other neurological diseases or psychological diseases
* Dementia
* Family history of epilepsy
* History of head trauma, surgery, or metal implants
* Having pacemaker or other electrical stimulators
* History of syncopes or frequent migraines

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Changes of transcranial magnetic stimulation (TMS) parameters | TMS parameters are assessed immediately before and after a 30-minute intervention. The data will be reported through study completion, for average of 6 months.
  Single-pulse and paired-pulse TMS are used to measure the cortical excitability of the motor cortex and the integrity of the intracortical inhibitory/facilitatory circuits. The TMS parameters include motor threshold (MT), motor evoke potential, silent period, short intracortical inhibition and facilitation. In single-pulse condition, the stimulation intensity is set at 130% of the MT. While in the paired-pulse condition, the first conditioning stimulus is set at 80% of MT, the second test stimulus is set at 130% of MT.

SECONDARY OUTCOMES:
Variation of walking step time | The step time variability is assessed immediately before and after a 30-minute intervention. The data will be reported through study completion, for average of 6 months.
  Subjects are asked to walk on a GAITRite carpet under usual walking speed. Duration between each step can be recorded through the system.
Walking ability | The walking ability is assessed immediately before and after a 30-minute intervention. The data will be reported through study completion, for average of 6 months.
  Walking speed, stride length and cadence are recorded as secondary outcome measures. Subjects are asked to walk on a GAITRite carpet under usual walking speed.
Variation of stepping-in-place movement | The step variability is assessed immediately before and after a 30-minute intervention. The data will be reported through study completion, for average of 6 months.
  Subjects are asked to stand and do stepping-in-place movement on a force plate.We use force plate to detect the vertical force and calculate the variation of each step.

CONTACTS AND LOCATIONS:
Overall Officials: Jau Yih Tsauo, PT, phD, Study Chair — department of physical therapy, college of medicine, National Taiwan University
Locations (1):
- Department of physical therapy, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No